CLINICAL TRIAL: NCT04373096
Title: Development of a Novel Hood Shield to Enhance PPE Security and Minimize COVID-19 Transmission to Front-line Health Care Workers Performing High-risk Procedures
Brief Title: Enhanced Hood PPE to Minimize COVID-19 Transmission to Front-line Health Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-5448
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-04

CONDITIONS: Covid19
Keywords: Enhanced PPE; Hood
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research coordinator documenting all outcome data will be blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Control) (Active Comparator): Will use current IPAC-UHN PPE as described under assigned intervention:
  Interventions: Device: current IPAC-UHN PPE
- Group H (enhanced PPE group ) (Experimental): Will use modified IPAC-UHN PPE including the prototype hood as described under assigned intervention:
  Interventions: Device: modified IPAC-UHN PPE

INTERVENTIONS:
Device: current IPAC-UHN PPE — * Fit-tested N95 mask
  * Open face shield
  * Double extended-cuff
  Arms: Group C (Control)
Device: modified IPAC-UHN PPE — * Fit-tested N95 mask
  * Hood
  * Double extended-cuff gloves
  Arms: Group H (enhanced PPE group )

SUMMARY:
This study proposes to compare the effectiveness of two different levels of PPE in protecting front-line health care workers from self-contamination with droplets and aerosolized particles during a simulated endotracheal intubation, an aerosol-generating medical procedure.

DETAILED DESCRIPTION:
Hospital acquired infection and death of healthcare workers is an alarming problem during the COVID-19 pandemic. Avoiding transmission of COVID-19 to front-line health care workers in Ontario with optimal Protective Personal Equipment (PPE) is a public health priority to prevent attrition of the health care work force at a time when it is most needed to care for the needs of Ontarians.

Health care workers performing Aerosol Generating Medical Procedures (AGMPs) (e.g. endotracheal intubation, bronchoscopy and tracheostomies) are at particularly high risk of infection. During AGMPs, medical personnel are contaminated with virus-loaded micro-droplets that may be suspended in the air for up to 3 hours.

Use of effective PPE is paramount in protecting health care workers during these high-risk procedures. Limited world-wide supplies of PPE and disruption of supply chains is a current concern. Having local sources of PPE production could help secure supply and protect Ontario's health care work force.

Current standard PPE equipment used during high-risk procedures in Ontario includes a fit-tested N95 mask, an open face shield, a procedure gown and double extended-cuff gloves. This level of PPE leaves certain areas of the head and neck exposed to contamination with viral aerosol and droplets, and could be a source for self-contamination despite meticulous donning and doffing. In fact, extensive contamination of the front surfaces, the neck, forearms, wrists and hands has been previously identified during simulation of medical procedures.

Contamination of the upper body, especially the head and neck, hands and wrists poses the highest risk of potential infection as viral contaminants in these parts of the body are most likely to reach the mucosal surfaces of the mouth, nose and eyes, which are the recognized entry points of viral infection.

The investigators propose to design and test a protective hood to be used in place of the open shield to provide enhanced coverage of the upper body during high risk procedures. This hood would be used along an N95 mask, procedure gown and double extended-cuff gloves, allowing for effective barrier protection against SARS-CoV-2 rich droplets and microdroplets by providing the physician with a barrier that covers his/her upper torso from contamination.

In partnership with 2 Ontario companies (MVF & Associates and Piedmont Plastics), the investigatorshave designed a hood to cover the entire upper body from the head down to the elbows. The hood is made of polypropylene spunbond nonwoven fabric, a waterproof, air permeable material and a polycarbonate visor.

The use of a hood could positively impact the safety of airway management and other AGMPs during the pandemic by reducing contamination of the upper body. The proposed study is important because it is the first one to evaluate the potential impact of a hood to enhance PPE. Ultimately, decreased levels of contamination by droplets may effectively reduce the risk of health care worker infection by SARS CoV2 virus after an AGMP such as endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, ASA 1-2 members of intubating team (staff anesthesiologists, fellows, anesthesia assistants, nurses) at the Toronto Western Hospital, University Health Network.
2. Age 20-75
3. Male or female

Exclusion Criteria:

a. Lack of a donning and doffing PPE training session at TWH in the last 6 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of contamination of any part of the base clothing or exposed skin of the upper body | 0-1 hour After doffing is complete
  Incidence of contamination of any part of the base clothing or exposed skin of the upper body (head or neck, forearms, arms, wrists, hands or torso)

SECONDARY OUTCOMES:
1) Number of body areas contaminated | 0-1 hour After doffing is complete
  For the purpose of this outcome, the body will be divided in the following 10 areas: a) face, b) hair or posterior aspect of the head, c) right side of the neck, d) left side of the neck, e) right arm or forearm, f) left arm or forearm, g) left wrist or hand, h) right wrist or hand, i) torso, j) right or left lower extremity.
2) Number of discrete areas of contamination of <1 cm2 and >1 cm2 | 0-1 hour After doffing is complete
  Number of discrete areas of contamination of <1 cm2 and >1 cm2
3) Visibility during the simulated procedure | 0-1 hour After doffing is complete
  Rated by each subject on an 11-point numeric rating scale from 0 (no visibility due to fogging or physical interference of the PPE, leading to inability to perform the required procedures) to 10 (perfect visibility, no fogging or physical interference with required tasks)
4) Ease of intubation procedures when wearing PPE | 0-1 hour After doffing is complete
  Assessed using an 11-point numeric rating scale from 0 = extremely difficult PPE made it impossible to intubate, to 10 = Absolutely no obstruction or difficulty added by the PPE
5) Ease of breathing while wearing PPE | 0-1 hour After doffing is complete
  Assessed using an 11-point numeric rating scale from 0=felt suffocated, needed to remove the PPE before completing the task to 10 = no difficulty breathing
6) Thermal comfort while wearing the PPE | 0-1 hour After doffing is complete
  Reported on an 11-point numeric rating scale from 0 = extremely hot, needed to remove the PPE before completing the tasks to 10= no discomfort due to temperature
7) Incidence of breaching of doffing procedures | 0-1 hour After doffing is complete
  Doffing violations will be documented and will be defined as performing a maneuver out of sequence, touching an item of clothing out of sequence, tearing an item of protective clothing, or touching any body part other than an item of protective clothing before performing hand hygiene.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD,FRCPC, Principal Investigator — Toronto Western Hospital , UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Leyva F, Perlas A, Chin KJ, Soheili M, Li Q, Huszti E, Chan V. A hood shield reduces postdoffing contamination during simulated COVID-19 airway management: an exploratory, simulation-based randomized study. Can J Anaesth. 2023 May;70(5):869-877. doi: 10.1007/s12630-023-02400-x. Epub 2023 Apr 5. PMID 37020172